CLINICAL TRIAL: NCT02148328
Title: A Phase 1, Double-blind, Active-controlled, Randomized Study in Healthy Adults to Evaluate Safety, Tolerability, and Immunogenicity of a Trivalent and Quadrivalent Cell-based Virosomal Subunit Influenza Vaccine
Brief Title: Safety, Tolerability, and Immunogenicity Study of a Cell-based Virosomal Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR104114; FLUCELLFLZ1003 (Other: Crucell Holland BV); 2014-000573-39 (EudraCT Number)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Influenza
Keywords: Healthy participants; Immunogenicity; Influenza; Prevention; Safety
MeSH Terms: conditions — Influenza, Human | interventions — Inflexal V

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Trivalent virosomal influenza vaccine (Experimental): Trivalent virosomal influenza vaccine will be administered intramuscularly (injection of a substance into a muscle) on Day 1 in healthy participants.
  Interventions: Biological: Trivalent virosomal influenza vaccine
- Commercial vaccine 1 (Active Comparator): Trivalent commercial virosomal influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Interventions: Biological: Commercial vaccine 1
- Quadrivalent virosomal influenza vaccine (Experimental): Quadrivalent virosomal influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Interventions: Biological: Quadrivalent virosomal influenza vaccine
- Commercial vaccine 2 (Active Comparator): Quadrivalent commercial influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Interventions: Biological: Commercial vaccine 2

INTERVENTIONS:
Biological: Trivalent virosomal influenza vaccine — Trivalent virosomal influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Other Names: Trivalent FluCell
  Arms: Trivalent virosomal influenza vaccine
Biological: Commercial vaccine 1 — Trivalent commercial virosomal influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Other Names: Inflexal V (trivalent)
  Arms: Commercial vaccine 1
Biological: Quadrivalent virosomal influenza vaccine — Quadrivalent virosomal influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Other Names: Quadrivalent FluCell
  Arms: Quadrivalent virosomal influenza vaccine
Biological: Commercial vaccine 2 — Quadrivalent commercial influenza vaccine will be administered intramuscularly on Day 1 in healthy participants.
  Other Names: Fluarix Tetra (quadrivalent)
  Arms: Commercial vaccine 2

SUMMARY:
The purpose of this study is to examine the safety and tolerability after administration of trivalent and quadrivalent cell-based virosomal influenza vaccine in healthy adults.

DETAILED DESCRIPTION:
This is a double-blind and randomized study in healthy adults. The duration of study will be approximately 90 days per participant. The study will include 4 visits: Day 1 (for vaccination), Day 4, Day 22 and day 90 (Follow-up visits). Safety and tolerability will be assessed by the rate of solicited, unsolicited, and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults
* Body Mass Index <= 30 kilogram per square meter (kg/m^2)
* Written informed consent

Exclusion Criteria:

* Vaccination with 2013/2014-seasonal influenza vaccine and/or receipt of any vaccine in the 4 weeks preceding receipt of study vaccine and/or any vaccination planned within 3 weeks from the study vaccine
* Diagnosis (by rapid test, performed at clinic/hospital laboratory) of laboratory-confirmed influenza in the 2013/2014 season
* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (greater than or equal to 38.0 celcius)
* Pregnancy as assessed by urine pregnancy test before vaccination, or lactation. Women of childbearing potential (that is, not surgically sterilized/hysterectomized or post-menopausal for more than 2 years) will be excluded if one of the following criteria is met: 1). Intention to become pregnant during the course of the study or to donate eggs (ova, oocytes) for the purposes of assisted reproduction 2). If heterosexually active, not using or not willing to continue using a medically reliable method of contraception for the entire study duration (up to 90 days). A medically reliable method of contraception includes oral contraceptive preparation (for example pills), hormonal implant, progestative injection, patch contraceptive formulation, an intrauterine device, concomitant use of barrier method and spermicide, or another method considered sufficiently reliable by the investigator in individual cases

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Solicited Local Adverse Events (AEs) | Up to Day 8
  The local AEs pain, erythema, and induration at the study vaccine injection site will be noted in the participant Diary from Day 1 to Day 8. The extent (largest diameter) of any redness or induration should be measured daily and recorded, along with any functional limitation of activity. Local AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of participants with Solicited Systemic Adverse Events (AEs) | Up to Day 8
  The solicited systemic AEs headache, fatigue, myalgia, malaise, and shivering/rigors will be noted in the participant Diary from Day 1 to Day 8. Fever (defined as body temperature greater than 38.0 Celsius) is another solicited systemic AE. Local AEs will be graded according to severity as mild (grade 1), moderate (grade 2), severe (grade 3) and potentially life threatening (grade 4).
Number of participants with Unsolicited Adverse Events (AEs) | Up to Day 22
  Unsolicited AEs are all AEs the participants are not specifically asked about in the participant Diary.
Number of participants with Serious Adverse Events (SAEs) | Up to Day 90
  The SAE is a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization or is a suspected transmission of any infectious agent via medicinal product.

SECONDARY OUTCOMES:
Number of Participants with Seroconversion | Day 22
  Number of participants with seroconversion will be the participants with a greater than or equal to (>=) 4-fold increase in hemagglutination inhibition (HI) antibody titer and a titer of >=1:40 at Day 22. HI against homologous strains will be measured with the HI test in serum.
Number of Participants with Seroprotection | Baseline and Day 22
  Number of participants with seroprotection is defined as number of participants with HI antibody >=1:40 at Day 22. HI against homologous strains will be measured with the HI test in serum.
Change From Baseline in Geometric Mean Titer (GMT) of HI antibodies | Baseline and Day 22
  GMT and increase in GMT of HI antibodies from Baseline to Day 22 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (4):
- Belgium (4):
  - Aalst
  - Ghent
  - Merksem
  - Wilrijk